CLINICAL TRIAL: NCT05849363
Title: A Prospective Study of Surgical Treatment Strategies for Goal B Type Basilar Invagination in China
Brief Title: A Prospective Study of Surgical Treatment Strategies for Goal B Type Basilar Invagination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XW-NS-GBTBI
Record Dates: First submitted 2022-10-09; First posted 2023-05-08 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-03

CONDITIONS: Basilar Invagination; Prospective Study; Surgical Outcome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior fossa decompression (Experimental): Posterior arch of atlas removal, reconstruction of cisterna magna, decompression of cerebellum, detection of magendie foramen.
  Interventions: Procedure: Posterior fossa decompression
- Posterior Compression-Distraction-Reduction-Fixation (Experimental): After subperiosteal dissection, the facet joint was exposed. A 2-mm joint "scraper" with sharp edge was inserted into the joint capsule and rotated to remove the articular cartilage. A blunt-edged rotating distractor was then inserted into the joint space, and the facet was sequentially opened with larger and larger blunt rotating distractors. After distraction on one side, an appropriate-sized trial was placed into the contralateral facet, holding the distraction open. This was repeated back and forth with larger trials. These steps were repeated, and the facet joints were distracted up to the pre-planned distance of the odontoid tip above Chamberlain's line.
  Interventions: Procedure: Posterior Compression-Distraction-Reduction-Fixation

INTERVENTIONS:
Procedure: Posterior fossa decompression — Posterior fossa decompression：Posterior arch of atlas removal, decompression of cerebellum, detection of foramen magnum.
  Arms: Posterior fossa decompression
Procedure: Posterior Compression-Distraction-Reduction-Fixation — Posterior Compression-Distraction-Reduction-Fixation：After subperiosteal dissection, the facet joint was exposed. A 2-mm joint "scraper" with sharp edge was inserted into the joint capsule and rotated to remove the articular cartilage. A blunt-edged rotating distractor was then inserted into the joint space, and the facet was sequentially opened with larger and larger blunt rotating distractors. After distraction on one side, an appropriate-sized trial was placed into the contralateral facet, holding the distraction open. This was repeated back and forth with larger trials. These steps were repeated, and the facet joints were distracted up to the pre-planned distance of the odontoid tip above Chamberlain's line.
  Arms: Posterior Compression-Distraction-Reduction-Fixation

SUMMARY:
The etiology of Goal B type basilar invagination (BI) is still not clear, and it may be related to platybasia and short slope. There is no unified standard surgical strategy for Goal B type BI, and different surgical strategies have a great influence on the surgical results of patients. The purpose of our prospective study in China is to (1) further clarify the etiology of Goal B type BI, and (2) improve the surgical outcome in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Goal B type basilar invagination (BI)

Exclusion Criteria:

* Preoperative diagnosis was confirmed as not Goal B type basilar invagination (BI)
* The patient was not physically fit for surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
JOA Score（Japanese Orthopaedic Association Scores） | 1 months, 3 months, and 6 months postoperatively
  Changes in JOA score，from 0 to 17, higher scores means better outcome
NDI Score | 1 months, 3 months, and 6 months postoperatively
  Changes in NDI score，from 0% to 100%，higher scores means worse outcome

SECONDARY OUTCOMES:
Change of Basilar Invagination | 1 months, 3 months, and 6 months postoperatively
  Radiographic assessment of the reduction of basilar invagination, using distance from odontoid tip to Chamberlain's line (DCL)
Change of CCA | 1 months, 3 months, and 6 months postoperatively
  Radiographic assessment of the change in clivus-canal angle (CCA)
Change of CVJ triangle area | 1 months, 3 months, and 6 months postoperatively
  Radiographic assessment of the reduction of CVJ triangle area
Change of CMA | 1 months, 3 months, and 6 months postoperatively
  Radiographic assessment of change of cervico-medullary angle (CMA)
Change of subarachnoid space | 1 months, 3 months, and 6 months postoperatively
  Radiographic assessment of the relief of width of subarachnoid space

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China